CLINICAL TRIAL: NCT01539538
Title: A Multicenter, Randomized, Open-Label, Parallel-Group Trial to Compare the Efficacy and Safety of the Sufentanil NanoTab PCA System/15 mcg (Zalviso™) to Intravenous Patient-Controlled Analgesia With Morphine for the Treatment of Acute Post-Operative Pain
Brief Title: A Multicenter, Randomized, Open-Label, Parallel-Group Trial to Compare the Efficacy and Safety of the Sufentanil NanoTab PCA System/15 mcg (Zalviso™)to Intravenous Patient-Controlled Analgesia With Morphine for the Treatment of Acute Post-Operative Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Talphera, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IAP309
Record Dates: First submitted 2012-02-22; First posted 2012-02-27 (Estimated); Results first posted 2014-03-27 (Estimated); Last update posted 2015-10-01 (Estimated); Status verified 2015-09

CONDITIONS: Post-Operative Pain
Keywords: Adult post-operative inpatients who; are expected to require parenteral; opioid analgesia for at least 48; hours after open abdominal surgery; or hip/knee replacement surgery
MeSH Terms: conditions — Pain, Postoperative | interventions — Sufentanil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sufentanil NanoTab PCA System/15 mcg (Experimental)
  Interventions: Drug: Sufentanil NanoTab PCA System/15 mcg
- morphine IV PCA (Active Comparator)
  Interventions: Drug: morphine IV PCA

INTERVENTIONS:
Drug: Sufentanil NanoTab PCA System/15 mcg — 15 mcg Sufentanil NanoTab dosed sublingually q 20 minutes as needed for pain for at least 48 hours and up to 72 hours
  Other Names: Zalviso™
  Arms: Sufentanil NanoTab PCA System/15 mcg
Drug: morphine IV PCA — 1 mg morphine administered IV q 6 minutes as needed for pain for at least 48 hours and up to 72 hours
  Arms: morphine IV PCA

SUMMARY:
The study is intended to show that the Sufentanil NanoTab PCA System is as effective as morphine intravenous patient-controlled analgesia (IV PCA) for treating pain after surgery. Each patient will use either the Sufentanil NanoTab PCA System or morphine IV PCA to treat their pain for at least 48 hours and up to 72 hours after surgery while in the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients who are 18 years or older
* Patients who are scheduled to undergo an open abdominal surgery (including laparoscopic-assisted), total knee or total hip replacement surgery under general anesthesia or spinal anesthesia that does not include intrathecal opioids during the operation.
* Post-surgical patients who have been admitted to the PACU and are expected to remain hospitalized and to have acute post-operative pain requiring parenteral opioids for at least 48 hours after surgery.

Exclusion Criteria:

* Patients who have taken an opioid for more than 30 consecutive days, at a daily dose of more than 15 mg of morphine (or equivalent), within the past 3 months prior to surgery (e.g. more than 3 doses per day of Vicodin®, Norco®, Lortab® with 5 mg hydrocodone per tablet).
* Patients with an allergy or hypersensitivity to opioids
* Female patients who are pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 357 (Actual)
Dates: Start 2012-04; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Palmer, M.D., PhD, Study Director — Talphera, Inc
Locations (16):
- United States (16):
  - Eliza Coffee Memorial Hospital, Florence, Alabama
  - Drug Research and Analysis Corp, Montgomery, Alabama
  - Shoals Medical Trials, Inc, Sheffield, Alabama
  - Arizona Research Center, Phoenix, Arizona
  - Lotus Clinical Research, Pasadena, California
  - Thorton Hospital, San Diego, California
  - Florida Research Associates, LLC, DeLand, Florida
  - River City Clinical Research, Jacksonville, Florida
  - Pensacola Research Consultants, Inc, Pensacola, Florida
  - Gulfcoast Research Institute, Sarasota, Florida
  - Phoenix Clinical Research LLC, Tamarac, Florida
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Access Clinical Trials, Nashville, Tennessee
  - Endeavor Clinical Trials, PA, San Antonio, Texas
  - Jean Brown Research, Salt Lake City, Utah

REFERENCES:
- [Background] Melson TI, Boyer DL, Minkowitz HS, Turan A, Chiang YK, Evashenk MA, Palmer PP. Sufentanil sublingual tablet system vs. intravenous patient-controlled analgesia with morphine for postoperative pain control: a randomized, active-comparator trial. Pain Pract. 2014 Nov;14(8):679-88. doi: 10.1111/papr.12238. Epub 2014 Aug 25. PMID 25155134

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sufentanil NanoTab PCA System/15 mcg | Morphine IV PCA
Started | 177 | 180
Completed | 146 | 136
Not Completed | 31 | 44
Not completed — Adverse Event | 13 | 18
Not completed — Lack of Efficacy | 13 | 16
Not completed — Withdrawal by Subject | 2 | 3
Not completed — PCA no longer required or PCA problem | 3 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sufentanil NanoTab PCA System/15 mcg | Morphine IV PCA | Total
Number analyzed (Participants) | 177 | 180 | 357
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 85 | 85 | 170
  >=65 years | 92 | 95 | 187
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (12.1) | 64 (12.6) | 64 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 123 | 108 | 231
  Male | 54 | 72 | 126
Region of Enrollment [Number; unit: participants]
  United States | 177 | 180 | 357

OUTCOME MEASURES:

1. Primary Outcome: Patient Global Satisfaction
Description: Proportion of patients responding good or excellent at 48-hour global assessment of method of pain control
Time Frame: 48 hours
Measure: Number (95% Confidence Interval); unit: % patients reporting good or excellent
Arm/Group | Sufentanil NanoTab PCA System/15 mcg | Morphine IV PCA
Number analyzed (Participants) | 177 | 180
% patients reporting good or excellent | 78.5 [72.5 to 84.6] | 65.6 [58.6 to 72.5]
Statistical Analysis 1: Comparison: Sufentanil NanoTab PCA System/15 mcg vs Morphine IV PCA; Test type: Non-Inferiority or Equivalence — Non-inferiority margin of - 15% for lower boundary of 95% confidence interval; p < 0.001, one-sided, z-test; difference in proportion = 12.90, 95% CI 2-sided [3.69 to 22.11]
Statistical Analysis 2: Comparison: Sufentanil NanoTab PCA System/15 mcg vs Morphine IV PCA; Test type: Superiority or Other; p = 0.007, t-test, 2 sided; Difference in proportion = 12.90

ADVERSE EVENTS:
Arm/Group | Sufentanil NanoTab PCA System/15 mcg | Morphine IV PCA
Serious Adverse Events (participants affected / at risk) | 6/177 | 7/180
Other Adverse Events (participants affected / at risk) | 123/177 | 122/180
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sufentanil NanoTab PCA System/15 mcg (N=177) | Morphine IV PCA (N=180)
post-procedural bile leak (Injury, poisoning and procedural complications) | 0 | 1
anaemia (Blood and lymphatic system disorders) | 1 | 1
methaemoglobinaemia (Blood and lymphatic system disorders) | 0 | 1
atrial fibrillation (Cardiac disorders) | 1 | 1
anastomotic haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
oxygen saturation decreased (Investigations) | 0 | 1
renal failure (Renal and urinary disorders) | 0 | 1
respiratory depression (Respiratory, thoracic and mediastinal disorders) | 1 | 0
haematoma (Vascular disorders) | 2 | 0
post-operative ileus (Injury, poisoning and procedural complications) | 1 | 0
hypotension (Vascular disorders) | 1 | 0
syncope (Nervous system disorders) | 1 | 0
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
ileus (Gastrointestinal disorders) | 0 | 1
anastomotic leak (Injury, poisoning and procedural complications) | 0 | 1
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
sepsis (Infections and infestations) | 0 | 1
abdominal distension (Gastrointestinal disorders) | 0 | 1
axillary vein thrombosis (Vascular disorders) | 1 | 0
clostridium difficile sepsis (Infections and infestations) | 1 | 0
peritonitis (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sufentanil NanoTab PCA System/15 mcg (N=177) | Morphine IV PCA (N=180)
nausea (Gastrointestinal disorders) | 76 | 72
vomiting (Gastrointestinal disorders) | 23 | 20
constipation (Gastrointestinal disorders) | 20 | 15
dyspepsia (Gastrointestinal disorders) | 6 | 2
oxygen saturation decreased (Investigations) | 17 | 17
headache (Nervous system disorders) | 14 | 12
dizziness (Nervous system disorders) | 10 | 6
confusional state (Psychiatric disorders) | 4 | 3
urinary retention (Renal and urinary disorders) | 2 | 5
pruritus (Skin and subcutaneous tissue disorders) | 7 | 14
hypotension (Vascular disorders) | 11 | 20
orthostatic hypotension (Vascular disorders) | 4 | 2
tachycardia (Cardiac disorders) | 2 | 3
bradycardia (Cardiac disorders) | 1 | 3 — All adverse events in this table were assessed by the PI as possibly or probably related to study drug
dry mouth (Gastrointestinal disorders) | 3 | 2
abdominal pain (Gastrointestinal disorders) | 0 | 3
abdominal distension (Gastrointestinal disorders) | 0 | 2
pyrexia (General disorders) | 2 | 3
procedural hypotension (Injury, poisoning and procedural complications) | 0 | 2
blood bilirubin increased (Investigations) | 1 | 2
hyponatremia (Metabolism and nutrition disorders) | 0 | 2
sedation (Nervous system disorders) | 2 | 1
somnolence (Nervous system disorders) | 1 | 2
insomnia (Psychiatric disorders) | 1 | 2
agitation (Psychiatric disorders) | 2 | 0
hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 2
hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
prior review and approval required